CLINICAL TRIAL: NCT00311311
Title: A Prospective, Randomized, Open-Label, Pilot Study To Compare The Effect On Carotid Atherosclerosis Of A Tacrolimus-Based Regimen With Conversion From A Tacrolimus- To A Sirolimus-Based Regimen At 3-4 Months Post-Transplant In De Novo Renal Transplant Recipients
Brief Title: Study Comparing Effect On Carotid Atherosclerosis Following Conversion From Tacrolimus To Sirolimus Post-Transplant In Kidney Transplant Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0468H1-319
Record Dates: First submitted 2006-04-03; First posted 2006-04-05 (Estimated); Results first posted 2012-05-24 (Estimated); Last update posted 2013-09-23 (Estimated); Status verified 2013-07

CONDITIONS: Atherosclerosis; Kidney Failure
Keywords: Kidney transplant; Renal transplant; Immunosuppression; Atherosclerosis; Graft Rejection
MeSH Terms: conditions — Atherosclerosis; Renal Insufficiency | interventions — Tacrolimus; Mycophenolic Acid; Prednisone; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Tacrolimus + MMF + Steroids
  Interventions: Drug: tacrolimus; Drug: mycophenolate mofetil; Drug: prednisone
- 2 (Experimental): Tacrolimus + MMF + Steroids with conversion from Tacrolimus to Sirolimus at 3-4 months post-transplant
  Interventions: Drug: sirolimus; Drug: tacrolimus; Drug: mycophenolate mofetil; Drug: prednisone

INTERVENTIONS:
Drug: tacrolimus — The daily dosage and formulation for each study treatment will be chosen by the investigator as medically appropriate for each individual subject, in order to achieve the target levels specified in the protocol TAC should be initiated within 24 hours before or after transplantation or within 14 days of transplantation as per local standard of care and tapered to a target trough level of 3-10 ng/mL by the Pre-Conversion visit at month 3-4 post-transplantation. The target trough level of TAC will be maintained at 3-10 ng/mL through to the end of the study.
  Other Names: CNI
  Arms: 1
Drug: mycophenolate mofetil — The daily dosage and formulation for each study treatment will be chosen by the investigator as medically appropriate for each individual subject, in order to achieve the target levels specified in the protocol MMF or MPS should be initiated within 24 hours before or after transplantation or within 14 days of transplantation per local standard of care and tapered to a minimum oral dose of MMF ≥ 500 mg/day or MPS ≥ 360 mg/day by the Pre-Conversion visit at month 3-4 post-transplantation. At the discretion of the investigator, MMF may be changed to MPS, or MPS may be changed to MMF. MMF is to be continued at ≥ 500 mg/day dose or MPS is to be continued at ≥ 360 mg/day dose through to the end of study.
  Other Names: MMF, MPS
  Arms: 1
Drug: prednisone — The daily dosage and formulation for each study treatment will be chosen by the investigator as medically appropriate for each individual subject, in order to achieve the target levels specified in the protocol CCS should be initiated within 24 hours before or after transplantation or within 14 days of transplantation per local standard of care and tapered to a minimum of 5 mg/day of prednisone orally or the alternate day equivalent by the Pre-Conversion visit at month 3-4 post-transplant. Continue administration of prednisone as per local standard of care to a minimum dose of 2.5 mg/day or alternate day equivalent dose to the end of the study. Withdrawal of CCS is prohibited.
  Other Names: CCS
  Arms: 1
Drug: sirolimus — The daily dosage and formulation for each study treatment will be chosen by the investigator as medically appropriate for each individual subject, in order to achieve the target levels specified in the protocol.
  On study Day 1 Conversion, the daily dose of TAC will not be taken, and SRL is initiated as a single 5-10 mg loading dose, followed by 3 mg/day on subsequent days, adjusted to maintain a SRL target trough level of 8-15 ng/mL through to month 24 post-transplant, then 5-12 ng/mL to the end of month 36 post-transplant.
  Arms: 2
Drug: tacrolimus — The daily dosage and formulation for each study treatment will be chosen by the investigator as medically appropriate for each individual subject, in order to achieve the target levels specified in the protocol TAC should be initiated within 24 hours before or after transplantation or within 14 days of transplantation as per local standard of care and tapered to a target trough level of 3-10 ng/mL by the Pre-Conversion visit at month 3-4 post-transplantation. Reintroduction of TAC or introduction of CsA is not permitted in the SRL Therapy group.
  Other Names: CNI
  Arms: 2
Drug: mycophenolate mofetil — The daily dosage and formulation for each study treatment will be chosen by the investigator as medically appropriate for each individual subject, in order to achieve the target levels specified in the protocol MMF or MPS should be initiated within 24 hours before or after transplantation or within 14 days of transplantation per local standard of care and tapered to a minimum oral dose of MMF ≥ 500 mg/day or MPS ≥ 360 mg/day by the Pre-Conversion visit at month 3-4 post-transplantation. At the discretion of the investigator, MMF may be changed to MPS, or MPS may be changed to MMF. MMF is to be continued at ≥ 500 mg/day dose or MPS is to be continued at ≥ 360 mg/day dose through to the end of study.
  Other Names: MMF, MPS
  Arms: 2
Drug: prednisone — The daily dosage and formulation for each study treatment will be chosen by the investigator as medically appropriate for each individual subject, in order to achieve the target levels specified in the protocol CCS should be initiated within 24 hours before or after transplantation or within 14 days of transplantation per local standard of care and tapered to a minimum of 5 mg/day of prednisone orally or the alternate day equivalent by the Pre-Conversion visit at month 3-4 post-transplant. Continue administration of prednisone as per local standard of care to a minimum dose of 2.5 mg/day or alternate day equivalent dose to the end of the study. Withdrawal of CCS is prohibited.
  Other Names: CCS
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether immunosuppression by tacrolimus, mycophenolate mofetil, and prednisone compared to conversion to sirolimus, mycophenolate mofetil, and prednisone affect the progression of atherosclerosis in renal transplant recipients.

DETAILED DESCRIPTION:
A decision to terminate the study was taken in November 2011 and a communication to that effect sent to all participating sites on November 18. All sites were asked to have patients returned to the sites and have all end of study procedures performed by Dec 31, 2011.

The decision to terminate this study was made following the conduct of an interim analysis which demonstrated that the study did not reach its primary endpoint. The termination of this study was not driven by any safety concerns and had no impact on subject safety and well-being.

ELIGIBILITY:
Inclusion Criteria:

At least one of the following characteristics:

* History of dialysis for at least 3 years.
* History of diabetes for at least 5 years.
* Hypertension or ischemic nephropathy as a cause of the end stage renal disease or loss of the first transplant.
* History of coronary artery disease, stroke, myocardial infarction, or amputation for vascular disease.

Exclusion Criteria:

* History of malignancy within the last 5 years (except adequately treated skin cancer).
* Recipients of non-renal organ transplant.
* Active gastrointestinal disease that may interfere with drug absorption.
* Active HIV, hepatitis B or C infection.
* Women who are pregnant or breastfeeding.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2006-04; Primary Completion 2010-12 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (7):
- Pfizer Investigational Site, Rochester, New York, United States
- Canada (6):
  - Pfizer Investigational Site, Calgary, Alberta
  - Pfizer Investigational Site, Edmonton, Alberta
  - Pfizer Investigational Site, Hamilton, Ontario
  - Pfizer Investigational Site, London, Ontario
  - Pfizer Investigational Site, Toronto, Ontario
  - Pfizer Investigational Site, Montreal, Quebec

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=0468H1-319&StudyName=Study%20Comparing%20Effect%20On%20Carotid%20Atherosclerosis%20Following%20Conversion%20From%20Tacrolimus%20To%20Sirolimus%20Post-Transplant%20In%20Kidney%20Transplant%20Pat

RESULTS

PARTICIPANT FLOW:
Groups:
- Tacrolimus Then Sirolimus With Mycophenolate/Prednisone: Participant received tacrolimus (TAC), (target trough level of 3-10 nanogram per milliliter [ng/mL] by 3-6 months post-transplant) plus mycophenolate mofetil (MMF) (greater than or equal to [>=] 500 milligram per day [mg/day]) or mycophenolate sodium (MPS) (>= 360 mg/day), plus prednisone (tapered to a minimum of 5 mg/day). Pre-randomization eligibility was assessed at Pre-Conversion Baseline (Weeks 12-24) and participants were randomized and assigned to treatment arm 0-14 days after Pre-Conversion Baseline. On Day 1 Conversion the participant stopped or tapered off TAC and began conversion to sirolimus (SRL- target trough level of 8-15 ng/mL through month 24 post-transplant and 5-12 ng/mL thereafter) + MMF (500-1500 mg/day) or MPS (360-1080 mg/day) or azathioprine (AZA) (50-75 mg/day) + prednisone (minimum of 2.5 mg/day) to end of study.
- Tacrolimus With Mycophenolate/Prednisone: Participant received TAC, target trough level of 3-10 ng/mL by 3-6 months post-transplant to end of study, plus MMF (>=500 mg/day) or MPS (>=360 mg/day) or AZA (>=50 mg/day) plus prednisone (>=2.5 mg/day), from day of transplant (Day 1) to end of study. TAC may have been converted to cyclosporine (CsA) (target CsA trough concentration [C0] level 50-250 ng/mL; target CsA concentration 2 hours post-dose [C2] level 200-1200 ng/mL) at the discretion of the investigator.
Period: Overall Study
Arm/Group | Tacrolimus Then Sirolimus With Mycophenolate/Prednisone | Tacrolimus With Mycophenolate/Prednisone
Started | 37 | 35
Completed | 29 | 26
Not Completed | 8 | 9
Not completed — Adverse Event | 3 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Noncompliance | 0 | 1
Not completed — Study Termination by Sponsor | 3 | 4
Not completed — Death | 1 | 0
Not completed — Lack of ancillary assistance | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Tacrolimus Then Sirolimus With Mycophenolate/Prednisone: Participant received tacrolimus (TAC), (target trough level of 3-10 ng/mL by 3-6 months post-transplant) plus MMF (>=500 mg/day) or mycophenolate sodium (MPS) (>=360 mg/day), plus prednisone (tapered to a minimum of 5 mg/day). Pre-randomization eligibility was assessed at Pre-Conversion Baseline (Weeks 12-24) and participants were randomized and assigned to treatment arm 0-14 days after Pre-Conversion Baseline. On Day 1 Conversion the participant stopped or tapered off TAC and began conversion to sirolimus (SRL- target trough level of 8-15 ng/mL through month 24 post-transplant and 5-12 ng/mL thereafter) + MMF (500-1500 mg/day) or MPS (360-1080 mg/day) or AZA (50-75 mg/day) + prednisone (minimum of 2.5 mg/day) to end of study.
- Tacrolimus With Mycophenolate/Prednisone: Participant received TAC, target trough level of 3-10 ng/mL by 3-6 months post-transplant to end of study, plus MMF (>=500 mg/day) or MPS (>=360 mg/day) or AZA (>=50 mg/day) plus prednisone (>=2.5 mg/day), from day of transplant (Day 1) to end of study. TAC may have been converted to CsA (target CsA trough concentration [C0] level 50-250 ng/mL; target CsA concentration 2 hours post-dose [C2] level 200-1200 ng/mL) at the discretion of the investigator.
- Total: Total of all reporting groups
Arm/Group | Tacrolimus Then Sirolimus With Mycophenolate/Prednisone | Tacrolimus With Mycophenolate/Prednisone | Total
Number analyzed (Participants) | 37 | 35 | 72
Age Continuous [Mean (Standard Deviation); unit: years] | 55.8 (11.11) | 55.5 (11.08) | 55.7 (11.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 9 | 20
  Male | 26 | 26 | 52

OUTCOME MEASURES:

1. Primary Outcome: Annual Change Rate in Total Plaque Volume (TPV) From Pre-conversion Baseline to 12 Months Post-transplant
Description: Within-subject annual change rate in TPV in the left and right distal common carotid arteries from the pre-conversion baseline to 12 months post kidney transplant as determined by ultrasound. Annual change rate equals (=) (TPV at month 12 post-transplant minus [-] TPV at pre-conversion baseline) divided (/) by imaging interval in years. TPV is the sum of assessment in left and right distal common carotid arteries.
Time Frame: Pre-conversion baseline and 12 months post-transplant
Population: On-Therapy Population: includes all intent-to-treat (ITT) subjects who also remained on assigned therapy until 12 months post-transplant for the primary endpoint, or until 36 months post-transplant for the cardiovascular and safety endpoints; N=number of evaluable participants for the outcome measure at 12 months post-transplant
Measure: Mean (Standard Deviation); unit: millimeter cube/year (mmˆ3/year)
Arm/Group | Tacrolimus Then Sirolimus With Mycophenolate/Prednisone | Tacrolimus With Mycophenolate/Prednisone
Number analyzed (Participants) | 18 | 20
millimeter cube/year (mmˆ3/year) | -49.31 (125.038) | 0.66 (23.103)

2. Primary Outcome: TPV at Pre-conversion Baseline
Description: TPV is the sum of the assessment in left and right distal common carotid arteries.
Time Frame: Pre-conversion baseline
Population: On-Therapy Population; N=number of evaluable participants for the outcome measure at pre-conversion Baseline
Measure: Mean (Standard Deviation); unit: mmˆ3
Arm/Group | Tacrolimus Then Sirolimus With Mycophenolate/Prednisone | Tacrolimus With Mycophenolate/Prednisone
Number analyzed (Participants) | 19 | 21
mmˆ3 | 68.68 (116.574) | 48.57 (72.207)

3. Secondary Outcome: Annual Change Rate in Carotid Intima Media Thickness (CIMT) From Pre-conversion Baseline at 12, 18, 24 and 36 Months Post-transplant
Description: Within-subject annual change rate in CIMT as determined by ultrasound. Mean CIMT=average of left CIMT and right CIMT. Annual CIMT Change Rate (mm/year) = (CIMT at Month x Post-transplant Visit - CIMT at Conversion Baseline) / Imaging interval in years.
Time Frame: Pre-conversion baseline, and 12, 18, 24 and 36 months post-transplant
Population: On-Therapy Population; N=number of evaluable participants; n=number of evaluable participants at specific time point
Measure: Mean (Standard Deviation); unit: millimeter/year (mm/year)
Arm/Group | Tacrolimus Then Sirolimus With Mycophenolate/Prednisone | Tacrolimus With Mycophenolate/Prednisone
Number analyzed (Participants) | 23 | 33
millimeter/year (mm/year)
  Annual Change Rate at 12 months (n=16,28) | 0.048 (0.0977) | 0.012 (0.0732)
  Annual Change Rate at 18 months (n=15,26) | 0.041 (0.0641) | -0.0002 (0.0543)
  Annual Change Rate at 24 months (n=15,23) | 0.023 (0.0614) | 0.015 (0.0453)
  Annual Change Rate at 36 months (n=8,13) | 0.028 (0.0381) | -0.007 (0.0460)
Statistical Analysis 1: Comparison: Tacrolimus Then Sirolimus With Mycophenolate/Prednisone vs Tacrolimus With Mycophenolate/Prednisone; 12 months post-transplant; Test type: Superiority or Other; p = 0.0445, ANCOVA — P-value and 95% CI for least square (LS) mean difference were calculated from repeated measures ANCOVA mixed model with baseline value, treatment group, time, and treatment group by time interaction as fixed effects, and subjects as random effect; Mean Difference (Final Values) = 0.036, 95% CI 2-sided [0.001 to 0.070] — LS mean difference
Statistical Analysis 2: Comparison: Tacrolimus Then Sirolimus With Mycophenolate/Prednisone vs Tacrolimus With Mycophenolate/Prednisone; 18 months post-transplant; Test type: Superiority or Other; p = 0.0288, ANCOVA — P-value and 95% CI for LS mean difference were calculated from repeated measures ANCOVA mixed model with baseline value, treatment group, time, and treatment group by time interaction as fixed effects, and subjects as random effect; Mean Difference (Final Values) = 0.034, 95% CI 2-sided [0.004 to 0.064] — LS mean difference
Statistical Analysis 3: Comparison: Tacrolimus Then Sirolimus With Mycophenolate/Prednisone vs Tacrolimus With Mycophenolate/Prednisone; 24 months post-transplant; Test type: Superiority or Other; p = 0.0269, ANCOVA — [p-value comment as in outcome 3, analysis 2]; Mean Difference (Final Values) = 0.032, 95% CI 2-sided [0.004 to 0.060] — LS mean difference
Statistical Analysis 4: Comparison: Tacrolimus Then Sirolimus With Mycophenolate/Prednisone vs Tacrolimus With Mycophenolate/Prednisone; 36 months post-transplant; Test type: Superiority or Other; p = 0.0970, ANCOVA — [p-value comment as in outcome 3, analysis 2]; Mean Difference (Final Values) = 0.028, 95% CI 2-sided [-0.005 to 0.060] — LS mean difference

4. Secondary Outcome: CIMT at Pre-conversion Baseline
Description: Mean CIMT=average of left CIMT and right CIMT.
Time Frame: Pre-conversion baseline
Population: On-Therapy Population; N=number of evaluable participants for the outcome measure at pre-conversion Baseline
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Tacrolimus Then Sirolimus With Mycophenolate/Prednisone | Tacrolimus With Mycophenolate/Prednisone
Number analyzed (Participants) | 17 | 29
mm | 0.735 (0.1502) | 0.773 (0.1391)

5. Secondary Outcome: Change From Pre-conversion Baseline in Carotid Plaque Roughness at 12 and 24 Months Post-transplant
Description: Carotid plaque roughness as determined by ultrasound. Change equals (=) value at post-transplant month x minus (-) pre-conversion baseline.
Time Frame: Pre-conversion baseline, 12, and 24 months post-transplant
Population: Evaluation of carotid plaque roughness at pre-conversion baseline, and at 12 and 24 months post-transplant was planned in the study design, however during the study conduct, it was removed as a cardiovascular endpoint since it was not validated.
Arm/Group | Tacrolimus Then Sirolimus With Mycophenolate/Prednisone | Tacrolimus With Mycophenolate/Prednisone
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change From Pre-conversion Baseline in Fasting Lipid Parameters at 12, 18, 24 and 36 Months Post-transplant
Description: Total Cholesterol (TC), Low Density Lipoprotein (LDL), High Density Lipoprotein (HDL) and Triglyceride (Tg) blood concentrations. Higher levels of TC, LDL and Tg are less desirable. Lower levels of HDL are less desirable. Change for each parameter = value at 12, 18, 24 and 36 months post-transplant - value at pre-conversion baseline.
Time Frame: Pre-conversion baseline, and 12, 18, 24 and 36 months post-transplant
Population: On-Therapy Population; N=number of evaluable participants; n=number of evaluable participants at specific time point
Measure: Mean (Standard Deviation); unit: millimole/liter (mmol/L)
Arm/Group | Tacrolimus Then Sirolimus With Mycophenolate/Prednisone | Tacrolimus With Mycophenolate/Prednisone
Number analyzed (Participants) | 23 | 33
millimole/liter (mmol/L)
  Change in TC 12 Months post-transplant (n=23,30) | 0.510 (1.0743) | -0.164 (0.8271)
  Change in LDL 12 Months post-transplant (n=21,30) | 0.277 (0.8282) | -0.056 (0.5612)
  Change in HDL 12 Months post-transplant (n=23,30) | 0.059 (0.3009) | -0.053 (0.4417)
  Change in Tg 12 Months post-transplant (n=23,30) | 0.617 (1.1135) | -0.117 (0.6088)
  Change in TC 18 Months post-transplant (n=21,29) | 0.361 (1.0704) | 0.082 (1.1427)
  Change in LDL 18 Months post-transplant (n=20,29) | 0.222 (0.9283) | 0.138 (0.8600)
  Change in HDL 18 Months post-transplant (n=21,29) | 0.106 (0.2824) | -0.030 (0.3601)
  Change in Tg 18 Months post-transplant (n=21,29) | 0.359 (0.9941) | -0.057 (0.8699)
  Change in TC 24 Months post-transplant (n=19,27) | 0.240 (1.1375) | -0.008 (1.0813)
  Change in LDL 24 Months post-transplant (n=16,27) | 0.067 (0.9493) | 0.054 (0.8250)
  Change in HDL 24 Months post-transplant (n=19,27) | 0.067 (0.2485) | -0.019 (0.3552)
  Change in Tg 24 Months post-transplant (n=19,27) | 0.547 (1.4083) | -0.088 (0.8131)
  Change in TC 36 Months post-transplant (n=15,21) | 0.386 (0.4841) | -0.323 (1.0652)
  Change in LDL 36 Months post-transplant (n=13,21) | 0.027 (0.5619) | -0.257 (0.8248)
  Change in HDL 36 Months post-transplant (n=15,21) | 0.098 (0.2141) | 0.111 (0.3042)
  Change in Tg 36 Months post-transplant (n=15,21) | 0.527 (0.9968) | -0.385 (0.7824)
Statistical Analysis 1: Comparison: Tacrolimus Then Sirolimus With Mycophenolate/Prednisone vs Tacrolimus With Mycophenolate/Prednisone; TC 12 Months Post-transplant; Test type: Superiority or Other; p < .0001, ANCOVA — P-value and 95% CI for LS mean difference were calculated from repeated measures ANCOVA mixed model with baseline value,treatment group,time and treatment group by time interaction as fixed effects,and subjects as random effect.ALPAH is unadjusted; Median Difference (Final Values) = 0.74, 95% CI 2-sided [0.39 to 1.09] — LS mean difference
Statistical Analysis 2: Comparison: Tacrolimus Then Sirolimus With Mycophenolate/Prednisone vs Tacrolimus With Mycophenolate/Prednisone; LDL 12 Months Post-transplant; Test type: Superiority or Other; p = 0.0022, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 0.41, 95% CI 2-sided [0.15 to 0.67] — LS mean difference
Statistical Analysis 3: Comparison: Tacrolimus Then Sirolimus With Mycophenolate/Prednisone vs Tacrolimus With Mycophenolate/Prednisone; HDL 12 Months Post-transplant; Test type: Superiority or Other; p = 0.1612, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 0.08, 95% CI 2-sided [-0.03 to 0.19] — LS mean difference
Statistical Analysis 4: Comparison: Tacrolimus Then Sirolimus With Mycophenolate/Prednisone vs Tacrolimus With Mycophenolate/Prednisone; Tg 12 Months Post-transplant; Test type: Superiority or Other; p = 0.0005, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 0.56, 95% CI 2-sided [0.26 to 0.86] — LS mean difference
Statistical Analysis 5: Comparison: Tacrolimus Then Sirolimus With Mycophenolate/Prednisone vs Tacrolimus With Mycophenolate/Prednisone; TC 18 Months Post-transplant; Test type: Superiority or Other; p = 0.0006, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 0.66, 95% CI 2-sided [0.30 to 1.02] — LS mean difference
Statistical Analysis 6: Comparison: Tacrolimus Then Sirolimus With Mycophenolate/Prednisone vs Tacrolimus With Mycophenolate/Prednisone; LDL 18 Months Post-transplant; Test type: Superiority or Other; p = 0.0126, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 0.34, 95% CI 2-sided [0.08 to 0.61] — LS mean difference
Statistical Analysis 7: Comparison: Tacrolimus Then Sirolimus With Mycophenolate/Prednisone vs Tacrolimus With Mycophenolate/Prednisone; HDL 18 Months Post-transplant; Test type: Superiority or Other; p = 0.2380, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 0.06, 95% CI 2-sided [-0.04 to 0.17] — LS mean difference
Statistical Analysis 8: Comparison: Tacrolimus Then Sirolimus With Mycophenolate/Prednisone vs Tacrolimus With Mycophenolate/Prednisone; Tg 18 Months Post-transplant; Test type: Superiority or Other; p = 0.0003, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 0.58, 95% CI 2-sided [0.27 to 0.88] — LS mean difference
Statistical Analysis 9: Comparison: Tacrolimus Then Sirolimus With Mycophenolate/Prednisone vs Tacrolimus With Mycophenolate/Prednisone; TC 24 Months Post-transplant; Test type: Superiority or Other; p = 0.0065, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 0.59, 95% CI 2-sided [0.17 to 1.00] — LS mean difference
Statistical Analysis 10: Comparison: Tacrolimus Then Sirolimus With Mycophenolate/Prednisone vs Tacrolimus With Mycophenolate/Prednisone; LDL 24 Months Post-transplant; Test type: Superiority or Other; p = 0.0845, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 0.28, 95% CI 2-sided [-0.04 to 0.60] — LS mean difference
Statistical Analysis 11: Comparison: Tacrolimus Then Sirolimus With Mycophenolate/Prednisone vs Tacrolimus With Mycophenolate/Prednisone; HDL 24 Months Post-transplant; Test type: Superiority or Other; p = 0.3742, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 0.05, 95% CI 2-sided [-0.06 to 0.16] — LS mean difference
Statistical Analysis 12: Comparison: Tacrolimus Then Sirolimus With Mycophenolate/Prednisone vs Tacrolimus With Mycophenolate/Prednisone; Tg 24 Months Post-transplant; Test type: Superiority or Other; p = 0.0006, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 0.59, 95% CI 2-sided [0.27 to 0.92] — LS mean difference
Statistical Analysis 13: Comparison: Tacrolimus Then Sirolimus With Mycophenolate/Prednisone vs Tacrolimus With Mycophenolate/Prednisone; TC 36 Months Post-transplant; Test type: Superiority or Other; p = 0.1488, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 0.44, 95% CI 2-sided [-0.16 to 1.03] — LS mean difference
Statistical Analysis 14: Comparison: Tacrolimus Then Sirolimus With Mycophenolate/Prednisone vs Tacrolimus With Mycophenolate/Prednisone; LDL 36 Months Post-transplant; Test type: Superiority or Other; p = 0.5460, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 0.14, 95% CI 2-sided [-0.33 to 0.62] — LS mean difference
Statistical Analysis 15: Comparison: Tacrolimus Then Sirolimus With Mycophenolate/Prednisone vs Tacrolimus With Mycophenolate/Prednisone; HDL 36 Months Post-transplant; Test type: Superiority or Other; p = 0.7511, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-0.12 to 0.16] — LS mean difference
Statistical Analysis 16: Comparison: Tacrolimus Then Sirolimus With Mycophenolate/Prednisone vs Tacrolimus With Mycophenolate/Prednisone; Tg 36 Months Post-transplant; Test type: Superiority or Other; p = 0.0048, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 0.63, 95% CI 2-sided [0.20 to 1.06] — LS mean difference

7. Secondary Outcome: Change From Pre-conversion Baseline in Glucose at Months 12, 24 and 36 Post-transplant
Description: Fasting plasma glucose. Change = value at month x post-transplant - pre-conversion baseline values.
Time Frame: Pre-conversion baseline, 12, 24 and 36 months post-transplant
Population: On-Therapy Population; N=number of evaluable participants; n=number of evaluable participants at specific time point
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Tacrolimus Then Sirolimus With Mycophenolate/Prednisone | Tacrolimus With Mycophenolate/Prednisone
Number analyzed (Participants) | 23 | 33
mmol/L
  Change at 12 Months post-transplant (n=23,33) | 0.606 (2.9461) | -0.083 (1.7377)
  Change at 24 Months post-transplant (n=19,31) | 0.832 (2.2068) | -0.076 (2.3982)
  Change at 36 Months post-transplant (n=14,22) | 0.686 (2.3559) | -0.214 (1.8239)
Statistical Analysis 1: Comparison: Tacrolimus Then Sirolimus With Mycophenolate/Prednisone vs Tacrolimus With Mycophenolate/Prednisone; 12 months post-transplant; Test type: Superiority or Other; p = 0.1757, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 0.78, 95% CI 2-sided [-0.36 to 1.91] — LS mean difference
Statistical Analysis 2: Comparison: Tacrolimus Then Sirolimus With Mycophenolate/Prednisone vs Tacrolimus With Mycophenolate/Prednisone; 24 months post-transplant; Test type: Superiority or Other; p = 0.0509, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 0.94, 95% CI 2-sided [-0.00 to 1.89] — LS mean difference
Statistical Analysis 3: Comparison: Tacrolimus Then Sirolimus With Mycophenolate/Prednisone vs Tacrolimus With Mycophenolate/Prednisone; 36 months post-transplant; Test type: Superiority or Other; p = 0.0683, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 1.11, 95% CI 2-sided [-0.09 to 2.31] — LS mean difference

8. Secondary Outcome: Change From Pre-conversion Baseline in Insulin at Months 12, 24, and 36 Post-transplant
Description: Fasting insulin. Change = value at month x post-transplant - pre-conversion baseline.
Time Frame: Pre-conversion baseline, 12, 24 and 36 months post-transplant
Population: On-Therapy Population; N=number of evaluable participants; n=number of evaluable participants at specific time point
Measure: Mean (Standard Deviation); unit: picomole/liter (pmol/L)
Arm/Group | Tacrolimus Then Sirolimus With Mycophenolate/Prednisone | Tacrolimus With Mycophenolate/Prednisone
Number analyzed (Participants) | 23 | 33
picomole/liter (pmol/L)
  Change at 12 Months post-transplant (n=16,23) | -4.549 (69.2139) | 17.953 (151.0513)
  Change at 24 Months post-transplant (n=13,23) | -6.120 (124.5500) | 32.180 (168.4674)
  Change at 36 Months post-transplant (n=10,14) | -22.759 (79.8717) | -2.731 (37.6576)
Statistical Analysis 1: Comparison: Tacrolimus Then Sirolimus With Mycophenolate/Prednisone vs Tacrolimus With Mycophenolate/Prednisone; 12 months post-transplant; Test type: Superiority or Other; p = 0.2741, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = -37.47, 95% CI 2-sided [-105.79 to 30.85] — LS mean difference
Statistical Analysis 2: Comparison: Tacrolimus Then Sirolimus With Mycophenolate/Prednisone vs Tacrolimus With Mycophenolate/Prednisone; 24 months post-transplant; Test type: Superiority or Other; p = 0.4865, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = -19.97, 95% CI 2-sided [-77.48 to 37.53] — LS mean difference
Statistical Analysis 3: Comparison: Tacrolimus Then Sirolimus With Mycophenolate/Prednisone vs Tacrolimus With Mycophenolate/Prednisone; 36 months post-transplant; Test type: Superiority or Other; p = 0.9339, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = -2.48, 95% CI 2-sided [-62.54 to 57.59] — LS mean difference

9. Secondary Outcome: Change From Pre-conversion Baseline in Glycosylated Hemoglobin(HbA1C) at Months 12, 24, and 36 Post-transplant
Description: HbA1C, change = value at month x post-transplant - pre-conversion baseline.
Time Frame: Pre-conversion baseline, 12, 24 and 36 months post-transplant
Population: On-Therapy Population; N=number of evaluable participants; n=number of evaluable participants at the specific time point
Measure: Mean (Standard Deviation); unit: percentage of glucose
Arm/Group | Tacrolimus Then Sirolimus With Mycophenolate/Prednisone | Tacrolimus With Mycophenolate/Prednisone
Number analyzed (Participants) | 23 | 33
percentage of glucose
  Change at 12 Months post-transplant (n=23,26) | 0.008 (0.0176) | 0.001 (0.0175)
  Change at 24 Months post-transplant (n=17,25) | 0.009 (0.0161) | 0.006 (0.0200)
  Change at 36 Months post-transplant (n=14,16) | 0.012 (0.0208) | -0.001 (0.0232)
Statistical Analysis 1: Comparison: Tacrolimus Then Sirolimus With Mycophenolate/Prednisone vs Tacrolimus With Mycophenolate/Prednisone; 12 months post-transplant; Test type: Superiority or Other; p = 0.4892, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 0.003, 95% CI 2-sided [-0.005 to 0.011] — LS mean difference
Statistical Analysis 2: Comparison: Tacrolimus Then Sirolimus With Mycophenolate/Prednisone vs Tacrolimus With Mycophenolate/Prednisone; 24 months post-transplant; Test type: Superiority or Other; p = 0.0514, ANCOVA — [p-value comment as in outcome 6, analysis 1]; LS mean difference; Mean Difference (Final Values) = 0.006, 95% CI 2-sided [-0.000 to 0.012]
Statistical Analysis 3: Comparison: Tacrolimus Then Sirolimus With Mycophenolate/Prednisone vs Tacrolimus With Mycophenolate/Prednisone; 36 months post-transplant; Test type: Superiority or Other; p = 0.1180, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 0.009, 95% CI 2-sided [-0.002 to 0.020] — LS mean difference

10. Secondary Outcome: Change From Pre-conversion Baseline in Adiponectin at Months 12, 24 and 36 Post-transplant
Description: Adiponectin is a biomarker for cardiovascular disease and atherosclerosis risk. A higher level indicates less risk. Change = month x post-transplant values - pre-conversion baseline values.
Time Frame: Pre-conversion baseline, 12, 24 and 36 months post-transplant
Population: On-Therapy Population; N=number of evaluable participants; n=number of evaluable participants at specific time point
Measure: Mean (Standard Deviation); unit: microgram per milliliter (µg/mL)
Arm/Group | Tacrolimus Then Sirolimus With Mycophenolate/Prednisone | Tacrolimus With Mycophenolate/Prednisone
Number analyzed (Participants) | 23 | 33
microgram per milliliter (µg/mL)
  Change at 12 Months post-transplant (n=23,33) | 5.352 (5.8935) | -2.205 (8.2503)
  Change at 24 Months post-transplant (n=18,31) | 2.244 (7.3628) | -0.267 (6.6144)
  Change at 36 Months post-transplant (n=15,22) | 1.487 (6.0933) | -1.413 (8.8053)
Statistical Analysis 1: Comparison: Tacrolimus Then Sirolimus With Mycophenolate/Prednisone vs Tacrolimus With Mycophenolate/Prednisone; 12 months post-transplant; Test type: Superiority or Other; p = 0.0016, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 5.56, 95% CI 2-sided [2.20 to 8.93] — LS mean difference
Statistical Analysis 2: Comparison: Tacrolimus Then Sirolimus With Mycophenolate/Prednisone vs Tacrolimus With Mycophenolate/Prednisone; 24 months post-transplant; Test type: Superiority or Other; p = 0.0091, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 3.91, 95% CI 2-sided [1.01 to 6.80] — LS mean difference
Statistical Analysis 3: Comparison: Tacrolimus Then Sirolimus With Mycophenolate/Prednisone vs Tacrolimus With Mycophenolate/Prednisone; 36 months post-transplant; Test type: Superiority or Other; p = 0.2468, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 2.25, 95% CI 2-sided [-1.60 to 6.10] — LS mean difference

11. Secondary Outcome: Change From Pre-conversion Baseline in High Sensitivity C-Reactive Protein (hsCRP) at Months 12, 24 and 36 Post-transplant.
Description: hsCRP is a biomarker of cardiovascular disease and atherosclerosis risk. A higher level indicates a greater risk. Change = month x post-transplant values - pre-conversion baseline values.
Time Frame: Pre-conversion baseline, 12, 24 and 36 months post-transplant
Population: On-Therapy Population; N=number of evaluable participants; n=number of evaluable participants at specific time point
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Tacrolimus Then Sirolimus With Mycophenolate/Prednisone | Tacrolimus With Mycophenolate/Prednisone
Number analyzed (Participants) | 23 | 33
mg/L
  Change at 12 Months post-transplant (n=23,33) | 1.611 (9.7219) | 1.379 (6.7680)
  Change at 24 Months post-transplant (n=18,31) | -0.563 (4.8347) | 1.723 (7.6259)
  Change at 36 Months post-transplant (n=15,22) | 0.336 (11.3537) | 3.164 (12.5660)
Statistical Analysis 1: Comparison: Tacrolimus Then Sirolimus With Mycophenolate/Prednisone vs Tacrolimus With Mycophenolate/Prednisone; 12 months post-transplant; Test type: Superiority or Other; p = 0.5282, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 0.95, 95% CI 2-sided [-2.05 to 3.94] — LS mean difference
Statistical Analysis 2: Comparison: Tacrolimus Then Sirolimus With Mycophenolate/Prednisone vs Tacrolimus With Mycophenolate/Prednisone; 24 months post-transplant; Test type: Superiority or Other; p = 0.5057, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 1.27, 95% CI 2-sided [-2.53 to 5.07] — LS mean difference
Statistical Analysis 3: Comparison: Tacrolimus Then Sirolimus With Mycophenolate/Prednisone vs Tacrolimus With Mycophenolate/Prednisone; 36 months post-transplant; Test type: Superiority or Other; p = 0.5701, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 1.59, 95% CI 2-sided [-4.00 to 7.18] — LS mean difference

12. Secondary Outcome: Change From Pre-conversion Baseline in Tumor Necrosis Factor Alpha (TNF-alpha) at Months 12, 24 and 36 Post-transplant
Description: TNF-alpha is a biomarker for cardiovascular disease and atherosclerosis risk. A higher level indicates a greater risk. Change = month x post-transplant values - pre-conversion baseline values.
Time Frame: Pre-conversion baseline, 12, 24 and 36 months post-transplant
Population: On-Therapy Population; N=number of evaluable participants; n=number of evaluable participants at specific time point
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Tacrolimus Then Sirolimus With Mycophenolate/Prednisone | Tacrolimus With Mycophenolate/Prednisone
Number analyzed (Participants) | 23 | 33
pg/mL
  Change at 12 Months post-transplant (n=23,32) | 0.991 (6.3462) | 0.000 (0.0000)
  Change at 24 Months post-transplant (n=18,30) | -0.367 (1.5580) | 1.894 (10.3720)
  Change at 36 Months post-transplant (n=15,22) | -0.441 (1.7067) | 0.000 (0.0000)

13. Secondary Outcome: Change From Pre-conversion Baseline in Endothelin-1 at Months 12, 24 and 36 Post-transplant
Description: Endothelin-1 is a biomarker for cardiovascular disease and atherosclerosis risk. A higher level indicates greater risk. Change = month x post-transplant values - pre-conversion baseline values.
Time Frame: Pre-conversion baseline, 12, 24 and 36 months post-transplant
Population: On-Therapy Population; N=number of evaluable participants; n=number of evaluable at the specific time point
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Tacrolimus Then Sirolimus With Mycophenolate/Prednisone | Tacrolimus With Mycophenolate/Prednisone
Number analyzed (Participants) | 23 | 33
pg/mL
  Change at 12 Months post-transplant (n=22,30) | 0.294 (0.4975) | 0.028 (0.4020)
  Change at 24 Months post-transplant (n=18,30) | 0.426 (0.5376) | 0.138 (0.8367)
  Change at 36 Months post-transplant (n=14,22) | 0.411 (0.7316) | -0.104 (0.7767)
Statistical Analysis 1: Comparison: Tacrolimus Then Sirolimus With Mycophenolate/Prednisone vs Tacrolimus With Mycophenolate/Prednisone; 12 months post-transplant; Test type: Superiority or Other; p = 0.0280, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 0.26, 95% CI 2-sided [0.03 to 0.48]
Statistical Analysis 2: Comparison: Tacrolimus Then Sirolimus With Mycophenolate/Prednisone vs Tacrolimus With Mycophenolate/Prednisone; 24 months post-transplant; Test type: Superiority or Other; p = 0.0190, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 0.26, 95% CI 2-sided [0.04 to 0.48]
Statistical Analysis 3: Comparison: Tacrolimus Then Sirolimus With Mycophenolate/Prednisone vs Tacrolimus With Mycophenolate/Prednisone; 36 months post-transplant; Test type: Superiority or Other; p = 0.1182, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 0.27, 95% CI 2-sided [-0.07 to 0.60]

14. Secondary Outcome: Change From Pre-conversion Baseline in Interleukin-6 (IL-6) at Months 12, 24 and 36 Post-transplant
Description: IL-6 is a biomarker for cardiovascular disease and atherosclerosis risk. A higher level indicates a greater risk. Change = month x post-transplant values - pre-conversion values.
Time Frame: Pre-conversion baseline, 12, 24 and 36 months post-transplant
Population: On-Therapy Population; N=number of evaluable participants; n=number of evaluable at the specific time point
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Tacrolimus Then Sirolimus With Mycophenolate/Prednisone | Tacrolimus With Mycophenolate/Prednisone
Number analyzed (Participants) | 23 | 33
pg/mL
  Change at 12 Months post-transplant (n=23,32) | -0.239 (3.6820) | 0.463 (3.8100)
  Change at 24 Months post-transplant (n=18,29) | 0.128 (6.9315) | 0.783 (4.7295)
  Change at 36 Months post-transplant (n=15,22) | -0.800 (3.8270) | 0.164 (6.4529)
Statistical Analysis 1: Comparison: Tacrolimus Then Sirolimus With Mycophenolate/Prednisone vs Tacrolimus With Mycophenolate/Prednisone; 12 months post-transplant; Test type: Superiority or Other; p = 0.7361, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = -0.30, 95% CI 2-sided [-2.09 to 1.49] — LS mean difference
Statistical Analysis 2: Comparison: Tacrolimus Then Sirolimus With Mycophenolate/Prednisone vs Tacrolimus With Mycophenolate/Prednisone; 24 months post-transplant; Test type: Superiority or Other; p = 0.5549, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = -0.53, 95% CI 2-sided [-2.32 to 1.26] — LS mean difference
Statistical Analysis 3: Comparison: Tacrolimus Then Sirolimus With Mycophenolate/Prednisone vs Tacrolimus With Mycophenolate/Prednisone; 36 months post-transplant; Test type: Superiority or Other; p = 0.6058, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = -0.76, 95% CI 2-sided [-3.69 to 2.17] — LS mean difference

15. Secondary Outcome: Change From Pre-conversion Baseline in Homocysteine at Months 12, 24 and 36 Post-transplant
Description: Homocysteine is a biomarker for cardiovascular disease and atherosclerosis risk. A higher level indicates a greater risk. Change = month x post-transplant values - pre-conversion baseline values.
Time Frame: Pre-conversion baseline, 12, 24 and 36 months post-transplant
Population: On-Therapy Population; N=number of evaluable participants; n=number of evaluable at the specific time point
Measure: Mean (Standard Deviation); unit: micromole/liter (µmol/L)
Arm/Group | Tacrolimus Then Sirolimus With Mycophenolate/Prednisone | Tacrolimus With Mycophenolate/Prednisone
Number analyzed (Participants) | 23 | 33
micromole/liter (µmol/L)
  Change at 12 Months post-transplant (n=23,33) | 1.278 (3.5572) | 0.530 (4.6244)
  Change at 24 Months post-transplant (n=19,31) | 1.316 (4.5373) | 2.158 (5.8978)
  Change at 36 Months post-transplant (n=15,22) | 1.087 (4.6641) | 2.459 (5.3116)
Statistical Analysis 1: Comparison: Tacrolimus Then Sirolimus With Mycophenolate/Prednisone vs Tacrolimus With Mycophenolate/Prednisone; 12 months post-transplant; Test type: Superiority or Other; p = 0.5902, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 0.60, 95% CI 2-sided [-1.63 to 2.84] — LS mean difference
Statistical Analysis 2: Comparison: Tacrolimus Then Sirolimus With Mycophenolate/Prednisone vs Tacrolimus With Mycophenolate/Prednisone; 24 months post-transplant; Test type: Superiority or Other; p = 0.7536, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = -0.36, 95% CI 2-sided [-2.68 to 1.95] — LS mean difference
Statistical Analysis 3: Comparison: Tacrolimus Then Sirolimus With Mycophenolate/Prednisone vs Tacrolimus With Mycophenolate/Prednisone; 36 months post-transplant; Test type: Superiority or Other; p = 0.4066, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = -1.33, 95% CI 2-sided [-4.53 to 1.86] — LS mean difference

16. Secondary Outcome: Change From Pre-conversion Baseline in Lipoprotein(a) at Months 12, 24 and 36 Post-transplant
Description: Lipoprotein(a) is a biomarker for cardiovascular disease and atherosclerosis risk. A higher level indicates a greater risk. Change = month x post-transplant values - pre-conversion baseline values.
Time Frame: Pre-conversion baseline, 12, 24 and 36 months post-transplant
Population: On-Therapy Population; N=number of evaluable participants; n=number of evaluable participants at specific time point
Measure: Mean (Standard Deviation); unit: milligram per deciliter (mg/dL)
Arm/Group | Tacrolimus Then Sirolimus With Mycophenolate/Prednisone | Tacrolimus With Mycophenolate/Prednisone
Number analyzed (Participants) | 23 | 33
milligram per deciliter (mg/dL)
  Change at 12 Months post-transplant (n=23,30) | 13.496 (23.3557) | -11.680 (77.1386)
  Change at 24 Months post-transplant (n=18,26) | 12.517 (36.8868) | 6.073 (31.5608)
  Change at 36 Months post-transplant (n=13,17) | 11.885 (49.4868) | 6.547 (22.0615)
Statistical Analysis 1: Comparison: Tacrolimus Then Sirolimus With Mycophenolate/Prednisone vs Tacrolimus With Mycophenolate/Prednisone; 12 months post-transplant; Test type: Superiority or Other; p = 0.3678, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 9.47, 95% CI 2-sided [-11.46 to 30.40] — LS mean difference
Statistical Analysis 2: Comparison: Tacrolimus Then Sirolimus With Mycophenolate/Prednisone vs Tacrolimus With Mycophenolate/Prednisone; 24 months post-transplant; Test type: Superiority or Other; p = 0.2179, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 10.72, 95% CI 2-sided [-6.53 to 27.97] — LS mean difference
Statistical Analysis 3: Comparison: Tacrolimus Then Sirolimus With Mycophenolate/Prednisone vs Tacrolimus With Mycophenolate/Prednisone; 36 months post-transplant; Test type: Superiority or Other; p = 0.3663, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 11.96, 95% CI 2-sided [-14.39 to 38.32] — LS mean difference

17. Secondary Outcome: Change From Pre-conversion Baseline in Fibrinogen at Months 12, 24 and 36 Post-transplant
Description: Fibrinogen is a biomarker for cardiovascular disease and atherosclerosis risk. A higher level indicates a greater risk. Change = month x post-transplant values - pre-conversion baseline values.
Time Frame: Pre-conversion baseline, 12, 24 and 36 months post-transplant
Population: On-Therapy Population; N=number of evaluable participants; n=number of evaluable participants at specific time point
Measure: Mean (Standard Deviation); unit: gram per liter (g/L)
Arm/Group | Tacrolimus Then Sirolimus With Mycophenolate/Prednisone | Tacrolimus With Mycophenolate/Prednisone
Number analyzed (Participants) | 23 | 33
gram per liter (g/L)
  Change at 12 Months post-transplant (n=22,31) | 0.62 (0.778) | 0.20 (0.769)
  Change at 24 Months post-transplant (n=19,29) | 0.45 (0.777) | 0.33 (0.741)
  Change at 36 Months post-transplant (n=14,20) | 0.40 (0.557) | 0.21 (0.740)
Statistical Analysis 1: Comparison: Tacrolimus Then Sirolimus With Mycophenolate/Prednisone vs Tacrolimus With Mycophenolate/Prednisone; 12 months post-transplant; Test type: Superiority or Other; p = 0.0410, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 0.4, 95% CI 2-sided [0.0 to 0.8] — LS mean difference
Statistical Analysis 2: Comparison: Tacrolimus Then Sirolimus With Mycophenolate/Prednisone vs Tacrolimus With Mycophenolate/Prednisone; 24 months post-transplant; Test type: Superiority or Other; p = 0.0275, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 0.3, 95% CI 2-sided [0.0 to 0.6] — LS mean difference
Statistical Analysis 3: Comparison: Tacrolimus Then Sirolimus With Mycophenolate/Prednisone vs Tacrolimus With Mycophenolate/Prednisone; 36 months post-transplant; Test type: Superiority or Other; p = 0.1841, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-0.1 to 0.6] — LS mean difference

18. Secondary Outcome: Change From Pre-conversion Baseline in Vitamin B12 at Months 12, 24 and 36 Post-transplant
Description: Vitamin B12 is a biomarker for cardiovascular disease and atherosclerosis risk. A lower level indicates a greater risk. Change = month x post-transplant values - pre-conversion values.
Time Frame: Pre-conversion baseline, 12, 24 and 36 months post-transplant
Population: On-Therapy Population; N=number of evaluable participants; n=number of evaluable participants at specific time points
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Tacrolimus Then Sirolimus With Mycophenolate/Prednisone | Tacrolimus With Mycophenolate/Prednisone
Number analyzed (Participants) | 23 | 33
pmol/L
  Change at 12 Months post-transplant (n=21,33) | -10.21 (161.662) | -11.38 (146.530)
  Change at 24 Months post-transplant (n=19,29) | -36.23 (88.910) | -27.46 (134.595)
  Change at 36 Months post-transplant (n=14,21) | -40.00 (135.353) | -46.39 (183.283)
Statistical Analysis 1: Comparison: Tacrolimus Then Sirolimus With Mycophenolate/Prednisone vs Tacrolimus With Mycophenolate/Prednisone; 12 months post-transplant; Test type: Superiority or Other; p = 0.0797, ANCOVA — [p-value comment as in outcome 6, analysis 1]; LS mean difference; Mean Difference (Final Values) = -51.3, 95% CI 2-sided [-108.9 to 6.3]
Statistical Analysis 2: Comparison: Tacrolimus Then Sirolimus With Mycophenolate/Prednisone vs Tacrolimus With Mycophenolate/Prednisone; 24 months post-transplant; Test type: Superiority or Other; p = 0.2341, ANCOVA — [p-value comment as in outcome 6, analysis 1]; LS mean difference; Mean Difference (Final Values) = -33.3, 95% CI 2-sided [-88.7 to 22.2]
Statistical Analysis 3: Comparison: Tacrolimus Then Sirolimus With Mycophenolate/Prednisone vs Tacrolimus With Mycophenolate/Prednisone; 36 months post-transplant; Test type: Superiority or Other; p = 0.6854, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = -15.2, 95% CI 2-sided [-90.3 to 59.8] — LS mean difference

19. Secondary Outcome: Change From Pre-conversion Baseline in Uric Acid at Months 12, 24 and 36 Post-transplant
Description: Uric Acid is a biomarker for cardiovascular disease and atherosclerosis risk. A higher level indicates a greater risk. Change = month x post-transplant values - pre-conversion baseline values.
Time Frame: Pre-conversion baseline, 12, 24 and 36 months post-transplant
Population: On-Therapy Population; N=number of evaluable participants; n=number of evaluable participants at specific time points
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | Tacrolimus Then Sirolimus With Mycophenolate/Prednisone | Tacrolimus With Mycophenolate/Prednisone
Number analyzed (Participants) | 23 | 33
µmol/L
  Change at 12 Months post-transplant (n=23,33) | -51.53 (68.987) | 11.10 (89.871)
  Change at 24 Months post-transplant (n=19,31) | -29.02 (93.350) | 3.89 (85.439)
  Change at 36 Months post-transplant (n=15,22) | -19.03 (83.162) | -0.58 (99.831)
Statistical Analysis 1: Comparison: Tacrolimus Then Sirolimus With Mycophenolate/Prednisone vs Tacrolimus With Mycophenolate/Prednisone; 12 months post-transplant; Test type: Superiority or Other; p = 0.0002, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = -72.8, 95% CI 2-sided [-108.6 to -36.9] — LS mean difference
Statistical Analysis 2: Comparison: Tacrolimus Then Sirolimus With Mycophenolate/Prednisone vs Tacrolimus With Mycophenolate/Prednisone; 24 months post-transplant; Test type: Superiority or Other; p = 0.0017, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = -67.6, 95% CI 2-sided [-108.5 to -26.6] — LS mean difference
Statistical Analysis 3: Comparison: Tacrolimus Then Sirolimus With Mycophenolate/Prednisone vs Tacrolimus With Mycophenolate/Prednisone; 36 months post-transplant; Test type: Superiority or Other; p = 0.0293, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = -62.3, 95% CI 2-sided [-118.2 to -6.5] — LS mean difference

20. Secondary Outcome: Change From Pre-conversion Baseline in Folate at 12, 24 and 36 Months Post-transplant
Description: Folate is a biomarker for cardiovascular disease and atherosclerosis risk. A lower level indicates a greater risk. Change = month x post-transplant values - pre-conversion baseline values.
Time Frame: Pre-conversion baseline, 12, 24 and 36 months post-transplant
Population: Two types of folate tests were used: serum folate and red blood cell (RBC) folate. The tests were not consistent across sites. Therefore, the evaluation was not analyzed.
Arm/Group | Tacrolimus Then Sirolimus With Mycophenolate/Prednisone | Tacrolimus With Mycophenolate/Prednisone
Number analyzed (Participants) | 0 | 0

21. Secondary Outcome: Number of Participants Who Used Lipid Lowering Therapies
Description: Participants who reported "yes" for taking lipid lowering therapies as concomitant medication.
Time Frame: From consent to conversion, from conversion to Month 12, from Months 12 to 24, and from Months 24 to 36 post-transplant
Population: On-Therapy Population; N=number of evaluable participants; n=number of evaluable at the specific time point
Measure: Number; unit: participants
Arm/Group | Tacrolimus Then Sirolimus With Mycophenolate/Prednisone | Tacrolimus With Mycophenolate/Prednisone
Number analyzed (Participants) | 23 | 33
participants
  From consent to conversion | 13 | 24
  From conversion to Month 12 | 22 | 29
  From Months 12 to Month 24 | 23 | 28
  From Months 24 to Month 36 | 18 | 27
Statistical Analysis 1: Comparison: Tacrolimus Then Sirolimus With Mycophenolate/Prednisone vs Tacrolimus With Mycophenolate/Prednisone; Use Lipid-Lowering From Consent to Conversion; Test type: Superiority or Other; p = 0.2573, Fisher Exact — P-value was calculated from 2-sided Fisher's exact test. Alpha is unadjusted
Statistical Analysis 2: Comparison: Tacrolimus Then Sirolimus With Mycophenolate/Prednisone vs Tacrolimus With Mycophenolate/Prednisone; Use Lipid-Lowering From Conversion to Month 12; Test type: Superiority or Other; p = 0.6386, Fisher Exact — P-value was calculated from 2-sided Fisher's exact test. Alpha is unadjusted
Statistical Analysis 3: Comparison: Tacrolimus Then Sirolimus With Mycophenolate/Prednisone vs Tacrolimus With Mycophenolate/Prednisone; Use Lipid-Lowering From Month 12 to Month 24; Test type: Superiority or Other; p = 0.0709, Fisher Exact — P-value was calculated from 2-sided Fisher's exact test. Alpha is unadjusted
Statistical Analysis 4: Comparison: Tacrolimus Then Sirolimus With Mycophenolate/Prednisone vs Tacrolimus With Mycophenolate/Prednisone; Use Lipid-Lowering From Month 24 to Month 36; Test type: Superiority or Other; p = 1.0000, Fisher Exact — P-value was calculated from 2-sided Fisher's exact test. Alpha is unadjusted

22. Secondary Outcome: Number of Participants Who Used Anti-hypertensive Medications
Description: Participants who reported "yes" for taking anti-hypertensive medications as concomitant medication.
Time Frame: From consent to conversion, from conversion to Month 12, from Months 12 to 24, and from Months 24 to 36 post-transplant
Population: On-Therapy Population; N=number of evaluable participants; n=number of evaluable at the specific time point
Measure: Number; unit: participants
Arm/Group | Tacrolimus Then Sirolimus With Mycophenolate/Prednisone | Tacrolimus With Mycophenolate/Prednisone
Number analyzed (Participants) | 23 | 33
participants
  From consent to conversion | 19 | 30
  From conversion to Month 12 | 21 | 30
  From Months 12 to Month 24 | 21 | 30
  From Months 24 to Month 36 | 18 | 28
Statistical Analysis 1: Comparison: Tacrolimus Then Sirolimus With Mycophenolate/Prednisone vs Tacrolimus With Mycophenolate/Prednisone; Use Anti-hypertension From Consent to Conversion; Test type: Superiority or Other; p = 0.4286, Fisher Exact — P-value was calculated from 2-sided Fisher's exact test. Alpha is unadjusted
Statistical Analysis 2: Comparison: Tacrolimus Then Sirolimus With Mycophenolate/Prednisone vs Tacrolimus With Mycophenolate/Prednisone; Use Anti-hypertension From Conversion to Month 12; Test type: Superiority or Other; p = 1.0000, Fisher Exact — P-value was calculated from 2-sided Fisher's exact test. Alpha is unadjusted
Statistical Analysis 3: Comparison: Tacrolimus Then Sirolimus With Mycophenolate/Prednisone vs Tacrolimus With Mycophenolate/Prednisone; Use Anti-hypertension From Month 12 to Month 24; Test type: Superiority or Other; p = 1.0000, Fisher Exact — P-value was calculated from 2-sided Fisher's exact test. Alpha is unadjusted
Statistical Analysis 4: Comparison: Tacrolimus Then Sirolimus With Mycophenolate/Prednisone vs Tacrolimus With Mycophenolate/Prednisone; Use Anti-hypertension From Month 24 to Month 36; Test type: Superiority or Other; p = 1.0000, Fisher Exact — P-value was calculated from 2-sided Fisher's exact test. Alpha is unadjusted

23. Secondary Outcome: Annual Rate of Change in TPV From Pre-conversion Baseline to 18, 24 and 36 Months Post Transplant
Description: Within-subject annual change rate in TPV in the left and right distal common carotid arteries from the pre-conversion baseline to 18, 24 and 36 months post kidney transplant as determined by ultrasound. Annual change rate equals (=) (TPV at month 18, 24 and 36 post-transplant minus [-] TPV at pre-conversion baseline) divided (/) by imaging interval in years. TPV is the sum of assessment in left and right distal common carotid arteries.
Time Frame: Pre-conversion baseline, and 18, 24 and 36 months post-transplant
Population: On-Therapy Population; N=number of evaluable participants; n=number of evaluable participants at specific time point
Measure: Mean (Standard Deviation); unit: mmˆ3/year
Arm/Group | Tacrolimus Then Sirolimus With Mycophenolate/Prednisone | Tacrolimus With Mycophenolate/Prednisone
Number analyzed (Participants) | 23 | 33
mmˆ3/year
  Month 18 post-transplant (n=12,12) | 17.15 (92.151) | 19.71 (44.734)
  Month 24 post-transplant (n=11,14) | 25.28 (67.393) | 9.10 (39.707)
  Month 36 post-transplant (n=7,11) | 6.62 (66.240) | 8.98 (25.505)
Statistical Analysis 1: Comparison: Tacrolimus Then Sirolimus With Mycophenolate/Prednisone vs Tacrolimus With Mycophenolate/Prednisone; 18 months post-transplant; Test type: Superiority or Other; p = 0.2718, ANCOVA — [p-value comment as in outcome 3, analysis 2]; Mean Difference (Final Values) = -18.0, 95% CI 2-sided [-50.7 to 14.7] — LS mean difference
Statistical Analysis 2: Comparison: Tacrolimus Then Sirolimus With Mycophenolate/Prednisone vs Tacrolimus With Mycophenolate/Prednisone; 24 months post-transplant; Test type: Superiority or Other; p = 0.2729, ANCOVA — [p-value comment as in outcome 3, analysis 2]; Mean Difference (Final Values) = -14.7, 95% CI 2-sided [-41.6 to 12.1] — LS mean difference
Statistical Analysis 3: Comparison: Tacrolimus Then Sirolimus With Mycophenolate/Prednisone vs Tacrolimus With Mycophenolate/Prednisone; 36 months post-transplant; Test type: Superiority or Other; p = 0.2902, ANCOVA — [p-value comment as in outcome 3, analysis 2]; Mean Difference (Final Values) = -8.2, 95% CI 2-sided [-23.8 to 7.3] — LS mean difference

ADVERSE EVENTS:
Time Frame: From post-conversion to the end of the study (Month 36 post-transplant)
Description: The same event may appear as both an adverse event (AE) and a serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Arm/Group | Tacrolimus Then Sirolimus With Mycophenolate/Prednisone | Tacrolimus With Mycophenolate/Prednisone
Serious Adverse Events (participants affected / at risk) | 17/37 | 21/35
Other Adverse Events (participants affected / at risk) | 36/37 | 33/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tacrolimus Then Sirolimus With Mycophenolate/Prednisone (N=37) | Tacrolimus With Mycophenolate/Prednisone (N=35)
CARCINOMA (General disorders) | 1 | 1
CELLULITIS (General disorders) | 0 | 2
CHEST PAIN (General disorders) | 1 | 1
FEVER (General disorders) | 0 | 1
HERNIA (General disorders) | 1 | 2
IMMUNE SYSTEM DISORDER (General disorders) | 2 | 2
INFECTION (General disorders) | 2 | 3
SEPSIS (General disorders) | 1 | 1
VIRAL INFECTION (General disorders) | 2 | 2
ARTERIOSCLEROSIS (Cardiac disorders) | 0 | 2
CORONARY ARTERY DISORDER (Cardiac disorders) | 1 | 0
EMBOLUS (Cardiac disorders) | 1 | 0
MYOCARDIAL INFARCT (Cardiac disorders) | 2 | 1
PERIPHERAL VASCULAR DISORDER (Cardiac disorders) | 1 | 0
THROMBOPHLEBITIS (Cardiac disorders) | 1 | 0
THROMBOSIS (Cardiac disorders) | 0 | 1
ESOPHAGITIS (Gastrointestinal disorders) | 0 | 1
GASTROINTESTINAL HEMORRHAGE (Gastrointestinal disorders) | 0 | 2
HEPATITIS (Gastrointestinal disorders) | 0 | 1
NAUSEA (Gastrointestinal disorders) | 0 | 1
VOMITING (Gastrointestinal disorders) | 0 | 2
LEUKOPENIA (Blood and lymphatic system disorders) | 1 | 1
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 | 1
HYPONATREMIA (Metabolism and nutrition disorders) | 0 | 1
BONE DISORDER (Musculoskeletal and connective tissue disorders) | 0 | 1
BONE NECROSIS (Musculoskeletal and connective tissue disorders) | 0 | 1
CEREBRAL ISCHEMIA (Nervous system disorders) | 0 | 1
NEUROPATHY (Nervous system disorders) | 0 | 1
PARAPLEGIA (Nervous system disorders) | 1 | 0
HEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PHARYNGITIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PNEUMONIA (Respiratory, thoracic and mediastinal disorders) | 1 | 2
SINUSITIS (Respiratory, thoracic and mediastinal disorders) | 0 | 2
ACUTE KIDNEY FAILURE (Renal and urinary disorders) | 0 | 2
KIDNEY FAILURE (Renal and urinary disorders) | 0 | 1
KIDNEY FUNCTION ABNORMAL (Renal and urinary disorders) | 0 | 2
PROSTATIC CARCINOMA (Renal and urinary disorders) | 1 | 0
PYELONEPHRITIS (Renal and urinary disorders) | 2 | 2
URINARY TRACT INFECTION (Renal and urinary disorders) | 1 | 2
ACCIDENTAL INJURY (General disorders) | 1 | 0
INFECTION BACTERIAL (General disorders) | 1 | 1
VASCULAR ANOMALY (Cardiac disorders) | 0 | 1
HYPOCALCEMIA (Metabolism and nutrition disorders) | 0 | 1
ARTHROSIS (Musculoskeletal and connective tissue disorders) | 0 | 1
OSTEOMYELITIS (Musculoskeletal and connective tissue disorders) | 0 | 1
SKIN CARCINOMA (Skin and subcutaneous tissue disorders) | 0 | 2
ANGINA PECTORIS (Cardiac disorders) | 0 | 2
ATRIAL FIBRILLATION (Cardiac disorders) | 0 | 1
Congestive Heart Failure (Cardiac disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tacrolimus Then Sirolimus With Mycophenolate/Prednisone (N=37) | Tacrolimus With Mycophenolate/Prednisone (N=35)
ABDOMINAL PAIN (General disorders) | 3 | 3
ACCIDENTAL INJURY (General disorders) | 9 | 5
ASTHENIA (General disorders) | 5 | 2
BACK PAIN (General disorders) | 4 | 7
CHEST PAIN (General disorders) | 5 | 1
FLU SYNDROME (General disorders) | 2 | 4
HEADACHE (General disorders) | 3 | 2
IMMUNE SYSTEM DISORDER (General disorders) | 3 | 1
INFECTION (General disorders) | 9 | 7
PAIN (General disorders) | 7 | 7
VIRAL INFECTION (General disorders) | 4 | 7
ARTERIOSCLEROSIS (Cardiac disorders) | 1 | 2
HYPERTENSION (Cardiac disorders) | 5 | 2
HYPOTENSION (Cardiac disorders) | 2 | 1
APHTHOUS STOMATITIS (Gastrointestinal disorders) | 2 | 0
CONSTIPATION (Gastrointestinal disorders) | 6 | 3
DIARRHEA (Gastrointestinal disorders) | 5 | 5
FLATULENCE (Gastrointestinal disorders) | 3 | 1
GASTROENTERITIS (Gastrointestinal disorders) | 1 | 2
NAUSEA (Gastrointestinal disorders) | 3 | 2
STOMATITIS (Gastrointestinal disorders) | 4 | 0
VOMITING (Gastrointestinal disorders) | 2 | 2
ANEMIA (Blood and lymphatic system disorders) | 4 | 7
LEUKOPENIA (Blood and lymphatic system disorders) | 6 | 2
AVITAMINOSIS (Metabolism and nutrition disorders) | 0 | 2
CREATININE INCREASED (Metabolism and nutrition disorders) | 1 | 7
DIABETES MELLITUS (Metabolism and nutrition disorders) | 5 | 3
EDEMA (Metabolism and nutrition disorders) | 3 | 2
GLUCOSE TOLERANCE DECREASED (Metabolism and nutrition disorders) | 2 | 0
HYPERCALCEMIA (Metabolism and nutrition disorders) | 2 | 5
HYPERCHOLESTEREMIA (Metabolism and nutrition disorders) | 9 | 2
HYPERLIPEMIA (Metabolism and nutrition disorders) | 14 | 5
PERIPHERAL EDEMA (Metabolism and nutrition disorders) | 13 | 6
WEIGHT GAIN (Metabolism and nutrition disorders) | 5 | 6
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 7 | 4
ARTHROSIS (Musculoskeletal and connective tissue disorders) | 2 | 0
BONE DISORDER (Musculoskeletal and connective tissue disorders) | 3 | 3
JOINT DISORDER (Musculoskeletal and connective tissue disorders) | 2 | 0
INSOMNIA (Nervous system disorders) | 2 | 3
PARESTHESIA (Nervous system disorders) | 3 | 3
COUGH INCREASED (Respiratory, thoracic and mediastinal disorders) | 3 | 3
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 3 | 3
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 2 | 0
PHARYNGITIS (Respiratory, thoracic and mediastinal disorders) | 7 | 6
RHINITIS (Respiratory, thoracic and mediastinal disorders) | 2 | 4
ACNE (Skin and subcutaneous tissue disorders) | 2 | 0
DRY SKIN (Skin and subcutaneous tissue disorders) | 2 | 2
HERPES ZOSTER (Skin and subcutaneous tissue disorders) | 3 | 1
PRURITUS (Skin and subcutaneous tissue disorders) | 3 | 2
RASH (Skin and subcutaneous tissue disorders) | 7 | 3
SKIN BENIGN NEOPLASM (Skin and subcutaneous tissue disorders) | 1 | 4
SKIN DISORDER (Skin and subcutaneous tissue disorders) | 4 | 1
SKIN HYPERTROPHY (Skin and subcutaneous tissue disorders) | 1 | 3
SWEATING (Skin and subcutaneous tissue disorders) | 2 | 1
CONJUNCTIVITIS (Eye disorders) | 0 | 2
ALBUMINURIA (Renal and urinary disorders) | 9 | 2
HEMATURIA (Renal and urinary disorders) | 5 | 4
URINARY TRACT INFECTION (Renal and urinary disorders) | 4 | 5
FEVER (General disorders) | 2 | 1
LAB TEST ABNORMAL (General disorders) | 2 | 1
DEEP THROMBOPHLEBITIS (Cardiac disorders) | 2 | 0
ANOREXIA (Gastrointestinal disorders) | 0 | 2
DYSPEPSIA (Gastrointestinal disorders) | 0 | 3
GASTROINTESTINAL DISORDER (Gastrointestinal disorders) | 2 | 1
PARATHYROID DISORDER (Endocrine disorders) | 1 | 2
POLYCYTHEMIA (Blood and lymphatic system disorders) | 1 | 3
HYPERKALEMIA (Metabolism and nutrition disorders) | 0 | 3
HYPOKALEMIA (Metabolism and nutrition disorders) | 3 | 0
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 | 2
ANXIETY (Nervous system disorders) | 1 | 2
DIZZINESS (Nervous system disorders) | 0 | 4
BRONCHITIS (Respiratory, thoracic and mediastinal disorders) | 1 | 2
HERPES SIMPLEX (Skin and subcutaneous tissue disorders) | 2 | 1
NAIL DISORDER (Skin and subcutaneous tissue disorders) | 2 | 1
SKIN ULCER (Skin and subcutaneous tissue disorders) | 0 | 2
DYSURIA (Renal and urinary disorders) | 0 | 2
UREMIA (Renal and urinary disorders) | 0 | 2
URINARY INCONTINENCE (Renal and urinary disorders) | 0 | 2
HEALING ABNORMAL (Metabolism and nutrition disorders) | 3 | 0
PNEUMONIA (Respiratory, thoracic and mediastinal disorders) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.